CLINICAL TRIAL: NCT05714644
Title: Community Collaboration to Advance Racial/Ethnic Equity in CRC Screening
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stand Up To Cancer (Other); University of California, Los Angeles (Other); Great Plains Tribal Leaders Health Board (Unknown)
Responsible Party: Principal Investigator, Jennifer S Haas, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2022P001678
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The Health Centers are randomized to FIT testing or Cologuard.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Mailed FIT Kit (Active Comparator): A FIT kit mailed to the patient's home
  Interventions: Other: FIT kit Screening Test
- Cologuard (Active Comparator): A Cologuard test mailed to the patient's home
  Interventions: Other: Cologuard Screening Test

INTERVENTIONS:
Other: FIT kit Screening Test — FIT kit mailed to the patient's home
  Arms: Mailed FIT Kit
Other: Cologuard Screening Test — Cologuard test mailed to the patient's home
  Arms: Cologuard

SUMMARY:
The goal of this pragmatic randomized clinical trial is to compare two colorectal (CRC) screening outreach approaches (FIT and Cologuard) in community health centers (CHC) in patients overdue for CRC screening. The main questions the project aims to answer are: What screening test has a higher completion rate? What screening test is more feasible and acceptable in a CHC setting? Patients will be sent a CRC screening test in the mail and will be asked to complete it at home and mail it back. Researchers will compare the completion rates for each screening test and will also look at the overall completion rate of both tests.

DETAILED DESCRIPTION:
This is a 3-year pragmatic trial with four levels of intervention, including system-, provider-, patient-, and community-level components at each of the CARES clinical sites. Health system components will include the development and implementation of a CRC screening registry and tracking database to systematically and actively track patients overdue for screening, screening test completion, and abnormal screening results. Data systems will be coupled with process re-design to improve clinical workflow for screening outreach. Providers will receive educational support through a training session about the importance of CRC screening, screening test options, population management, and an instructional on how to complete a Cologuard kit (Cologuard arm only) or a FIT kit (FIT arm only). Patient components of the intervention vary by study arm. In sites randomized to Cologuard, patients will receive a mailed Cologuard kit and the Exact Sciences patient support program. Patients in clinics randomized to FIT will receive a mailed FIT kit with systematic reminders. Patients who test positive will be offered patient navigation to assist with completing a diagnostic colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75
2. Has had a visit at a participating community clinic within the last two years.
3. Alive
4. Patient's preferred language is English or Spanish

Exclusion Criteria:

Exclusion Criteria:

1. Has Ulcerative Colitis or Crohn's disease documented in the problem list. (Codes below).
2. Has colorectal cancer documented in the problem list. (Codes below).
3. Has had a FIT in the past 1 year
4. Has had a colonoscopy in the past 10 years

ICD-10 codes for exclusion criteria:

Ulcerative colitis:

* K51.0
* K51.2
* K51.3
* K51.4
* K51.5
* K51.8
* K51.9
* K52.8
* K52.9

Crohn's disease:

* K50.0
* K50.1
* K50.8
* K50.9

Colorectal cancer

* C18 (malignant neoplasm of colon)
* C18.0 (malignant neoplasm of cecum)
* C18.1 (malignant neoplasm of appendix)
* C18.2 (malignant neoplasm of ascending colon)
* C18.3 (malignant neoplasm of hepatic flexure)
* C18.4 (malignant neoplasm of transverse colon)
* C18.5 (malignant neoplasm of splenic flexure)
* C18.6 (malignant neoplasm of descending colon)
* C18.7 (malignant neoplasm of sigmoid colon)
* C18.8 (malignant neoplasm of overlapping sites of colon)
* C18.9 (malignant neoplasm of colon, unspecified)
* C19 (malignant neoplasm of rectosigmoid junction)
* C20 (malignant neoplasm of rectum)
* C21.8 (malignant neoplasm of overlapping sites of rectum, anus and anal canal)
* C26.0 (malignant neoplasm of intestinal tract, part unspecified)
* C78.5 (secondary malignant neoplasm of large intestine and rectum)
* C78.6 (secondary malignant neoplasm of retroperitoneum and peritoneum)
* D37.4 (neoplasm of uncertain behavior of colon)
* D37.5 (neoplasm of uncertain behavior of rectum)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5127 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Haas, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - UCLA, Los Angeles, California
  - Mass General Brigham, Boston, Massachusetts
  - Great Plains Tribal Leaders Health Board, Rapid City, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] May FP, Brodney S, Tuan JJ, Syngal S, Chan AT, Glenn B, Johnson G, Chang Y, Drew DA, Moy B, Rodriguez NJ, Warner ET, Anyane-Yeboa A, Ukaegbu C, Davis AQ, Schoolcraft K, Regan S, Yoguez N, Kuney S, Le Beaux K, Jeffries C, Lee ET, Bhat R, Haas JS. Community Collaboration to Advance Racial/Ethnic Equity in Colorectal Cancer Screening: Protocol for a Multilevel Intervention to Improve Screening and Follow-up in Community Health Centers. Contemp Clin Trials. 2024 Oct;145:107639. doi: 10.1016/j.cct.2024.107639. Epub 2024 Jul 26. PMID 39068985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Dates: 6/7/23 through 10/24/23
Pre-assignment Details: No enrolled patients were excluded from the study before assignment to arms.
Units Other Than Participants: community health center
Period: Overall Study
Arm/Group | Mailed FIT Kit | Cologuard
Started | 2435; 4 community health center | 2692; 4 community health center
Completed | 2435; 4 community health center | 2692; 4 community health center
Not Completed | 0; 0 community health center | 0; 0 community health center

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mailed FIT Kit | Cologuard | Total
Number analyzed (Participants) | 2435 | 2692 | 5127
Age, Continuous [Mean (Standard Deviation); unit: years] — Age
  years | 54.9 (8.1) | 54.2 (8.1) | 54.5 (8.1)
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity Population: Race/Ethnicity
  Participants
    Non-Hispanic, White | 456 | 307 | 763
    Non-Hispanic, Black | 196 | 173 | 369
    Hispanic | 1722 | 2096 | 3818
    Other/Unknown | 61 | 116 | 177
Sex: Female, Male [Count of Participants; unit: Participants] — Sex Population: Sex
  Participants
    Female | 1437 | 1581 | 3018
    Male | 998 | 1111 | 2109

OUTCOME MEASURES:

1. Primary Outcome: CRC Screening Completion Rates
Description: completion rate of the stool-based screening test (FIT or Cologuard)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mailed FIT Kit | Cologuard
Number analyzed (Participants) | 2435 | 2692
Participants | 550 | 751
Statistical Analysis 1: Comparison: Mailed FIT Kit vs Cologuard; Test type: Superiority — FIT-DNA hypothesized to be higher than FIT; p = 0.05, Regression, Logistic; logistic regression models with generalized estimating equations to account for clustering of data within CHCs, adjusting for age and race/ethnicity; Risk Difference (RD) = 4.7, 95% CI 2-sided [0.8 to 8.7]

2. Secondary Outcome: CRC Screening Completion Rates
Description: completion rate of the stool-based screening test (Cologuard or FIT)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mailed FIT Kit | Cologuard
Number analyzed (Participants) | 2435 | 2692
Participants | 649 | 854
Statistical Analysis 1: Comparison: Mailed FIT Kit vs Cologuard; Test type: Superiority — FIT-DNA greater than FIT; p < 0.05, Regression, Logistic; Risk Difference (RD) = 4.5, 95% CI 2-sided [0.4 to 8.5]

3. Secondary Outcome: Diagnostic Colonoscopy Completion Rates
Description: completion rate of diagnostic colonoscopy after an abnormal stool test result (overall and by arm)
Time Frame: 6 months
Population: The number is for participants who returned an abnormal stool test within 180 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Mailed FIT Kit | Cologuard
Number analyzed (Participants) | 42 | 58
Participants | 13 | 23

ADVERSE EVENTS:
Time Frame: From enrollment through 180 days for negative test result or an additional 180 days after a positive FIT or Cologuard was returned, up to 1 year.
Arm/Group | Mailed FIT Kit | Cologuard
All-Cause Mortality (participants affected / at risk) | 0/2435 | 0/2692
Serious Adverse Events (participants affected / at risk) | 0/2435 | 0/2692
Other Adverse Events (participants affected / at risk) | 0/2435 | 0/2692

LIMITATIONS AND CAVEATS:
Boston and LA used different FIT kit brands. No access to patient-level data about outreach attempts or contacts from the Exact Science patient support program because this information is proprietary.

Unable to comment on cost-effectiveness. Unable to randomize the South Dakota site because unable to identify another CHC in the region to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-10-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT05714644/Prot_003.pdf
  • Statistical Analysis Plan (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT05714644/SAP_004.pdf